CLINICAL TRIAL: NCT02030041
Title: Effect of Vitamin D Supplementation on Exercise Adaptations in Patients on Statin Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Ashu Rastogi, Asst Professor, Department of Endocrinology, Postgraduate Institute of Medical Education and Research, Chandigarh, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Simvavitd
Record Dates: First submitted 2013-12-23; First posted 2014-01-08 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-03-31 (Actual); Status verified 2017-02

CONDITIONS: Dyslipidemias
Keywords: simvastatin; cardiorespiratory fitness; vitamin D; exercise; mitochondria
MeSH Terms: conditions — Dyslipidemias; Motor Activity | interventions — Vitamin D; Cholecalciferol; Simvastatin; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Simvastatin and placebo (Experimental): Eleven participants will be vitamin D deficient with LDL-C between 100 to 130mg/dl.
  This arm will receive Simvastatin 40 mg once daily and placebo once weekly, and will perform moderate intensity exercise for twelve weeks. Participants will be advised to walk a minimum of 3000 steps in 30 minutes on 5 days each week
  Interventions: Drug: Simvastatin; Drug: Placebo
- Simvastatin and vitamin D (Active Comparator): Eleven participants will be vitaminD deficient with LDL-C between 100 to 130mg/dl.
  This arm will receive simvastatin 40 mg once daily and vitaminD 60,000 units once weekly , and will perform moderate intensity exercise for twelve weeks. Participants will be advised to walk a minimum of 3000 steps in 30 minutes on 5 days each week
  Interventions: Drug: Vitamin D; Drug: Simvastatin
- Vitamin D and placebo (Active Comparator): Eleven participants will be vitamin D deficient with LDL-C between 100 to 130mg/dl This arm will receive vitamin D 60,000 units once weekly and placebo once daily, and will perform moderate intensity exercise for twelve weeks. Participants will be advised to walk a minimum of 3000 steps in 30 minutes on 5 days each week
  Interventions: Drug: Vitamin D; Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D — Vitamin D will be given to achieve normal serum levels
  Other Names: Cholecalciferol
  Arms: Simvastatin and vitamin D; Vitamin D and placebo
Drug: Simvastatin — Simvastatin in a dose of 40 mg will be provided to the study participants
  Other Names: Statin
  Arms: Simvastatin and placebo; Simvastatin and vitamin D
Drug: Placebo — Placebo will be provided to the study participants
  Arms: Simvastatin and placebo; Vitamin D and placebo

SUMMARY:
Statins along with lifestyle modifications including exercise are commonly prescribed to patients with type 2 diabetes. American diabetes association recommends using moderate-intensity statin and lifestyle therapy for patients with diabetes aged ≥40 years, even without additional cardiovascular disease(CVD) risk factors.. Myopathy is a well known adverse effect of statins, which occurs in 1-7% of patients. The spectrum of statin-related myopathy ranges from common benign myalgia to rare but life threatening rhabdomyolysis. Being lipophilic, simvastatin diffuses nonselectively into extrahepatic tissues such as muscle, leading to higher incidence of myopathy among statin users.

In addition, simvastatin attenuates the exercise-induced increase in cardiorespiratory fitness, and reduces the skeletal muscle mitochondrial content and oxidative capacity in humans. Impaired cardiorespiratory fitness and mitochondrial function is possibly due to reduction in Coenzyme Q10, which is a component of the electron transport chain and is indispensable for generation of adenosine triphosphate (ATP) during oxidative phosphorylation in mitochondria. Statins or hydroxyl-methylglutaryl coenzyme A (HMA CoA) reductase inhibitors interfere with the production of mevalonic acid, which is a precursor in the synthesis of coenzyme Q10.

Mitochondrial dysfunction has also been reported in vitamin D deficient individuals which has been attributed to intra-mitochondrial calcium deficiency or deficient enzyme function of the oxidative pathway ( by direct effect of vitamin D on enzyme gene or protein expression). Thus, vitamin D may improve the statin-mediated changes in cardiorespiratory fitness and mitochondrial function by improving the enzymatic machinery involved in oxidative phosphorylation which is blocked by statin. This study is being done to look for the effect of vitamin D supplementation on simvastatin-mediated change in exercise-mediated cardiorespiratory fitness and skeletal muscle mitochondrial content in adults with type 2 diabetes

DETAILED DESCRIPTION:
Statins, a class of hydroxyl methylglutaryl-coenzyme A reductase inhibitors that lower low-density lipoprotein cholesterol, are commonly prescribed to patients with the metabolic syndrome or those with multiple cardiovascular disease risk factors when lifestyle changes fail to achieve LDL targets to reduce the risk of coronary heart disease morbidity and mortality. American Diabetes Association (ADA) recommends moderate intensity statin for patients with diabetes without additional CVD risk factors aged >40.Statins are widely prescribed in combination with exercise to lower risk of cardiovascular disease morbidity and mortality. Every 1millimole per liter reduction in LDL is associated with a 10-20% reduction in risk of cardiovascular events and all-cause mortality, while every 1 Metabolic equivalent [MET] (3.5 milliliters of oxygen per kilogram of body weight per minute) increase in fitness is associated with an 18% reduction in cardiovascular disease mortality and an 11-50% reduction in all-cause mortality.Statins are generally safe, but myotoxicity, including fatal rhabdomyolysis can occur. Although severe muscle-related side effects occur in <0.1% of statin users, less severe symptoms, such as myalgia and muscle cramps, occur in 1-7% of users.

The mechanisms mediating statin myopathy are unclear, but possibilities include decreased sarcolemmal or endoplasmic reticulum cholesterol, reduced production of prenylated proteins including the mitochondrial electron transport protein coenzyme Q10, reduced fat catabolism, increased myocellular concentrations of cholesterol and plant sterols, failure to repair damaged skeletal muscle, vitamin D deficiency, and inflammation. Increasingly, interest has focused on altered cellular energy use and mitochondrial dysfunction, with the dysfunction activating pathways leading to muscle atrophy. Although the mechanisms are poorly understood, some statins (simvastatin, atorvastatin, fluvastatin) have been shown to reduce skeletal muscle mitochondrial content and oxidative capacity in humans.

Sirvent et al evaluated the mitochondrial function and calcium signaling in muscles of patients treated with statins, who present or not muscle symptoms, by oxygraphy and recording of calcium sparks, respectively. Patients treated with statins showed impairment of mitochondrial respiration that involved mainly the complex I of the respiratory chain and altered frequency and amplitude of calcium sparks. The muscle problems observed in statin-treated patients appear thus to be related to impairment of mitochondrial function and muscle calcium homeostasis.

Mikus et al examined the effects of simvastatin on changes in cardiorespiratory fitness and skeletal muscle mitochondrial content in response to aerobic exercise training. The primary outcomes were cardiorespiratory fitness and skeletal muscle (vastus lateralis) mitochondrial content (citrate synthase enzyme activity). Thirty-seven participants (exercise plus statins; n=18; exercise only; n=19) completed the study. Cardiorespiratory fitness increased by 10% (P<0.05) in response to exercise training alone, but was blunted by the addition of simvastatin resulting in only a 1.5% increase (P<0.005 for group by time interaction). Similarly, skeletal muscle citrate synthase activity increased by 13% in the exercise only group (P <0.05), but decreased by 4.5% in the simvastatin plus exercise group (P<0.05 ) Impaired cardiorespiratory fitness and mitochondrial function is possibly due to reduction in Coenzyme Q10, which is a component of the electron transport chain and is indispensable for generation of ATP during oxidative phosphorylation in mitochondria. Statins or hydroxyl-methylglutaryl coenzyme A (HMA CoA) reductase inhibitors interfere with the production of mevalonic acid, which is a precursor in the synthesis of coenzyme Q10.

Mitochondrial dysfunction has also been reported in vitamin D deficient individuals which has been attributed to intra-mitochondrial calcium deficiency or deficient enzyme function of the oxidative pathway ( by direct effect of vitamin D on enzyme gene or protein expression).

Mukherjee et al conducted a study in which chicks were raised for 3 to 4 weeks either on a normal (vitamin D supplemented) or a rachitogenic diet. The Ca2+ content of the serum, heart tissue and heart mitochondria was significantly decreased in chicks raised on a rachitogenic diet. In mitochondria isolated from calcium deficient hearts, the rate of adenosine diphosphate induced state 3 respiration and 2,4-Dinitrophenol uncoupled respiration were significantly decreased.When vitamin D deficient chicks were orally dosed with vitamin D3, serum calcium level and state 3 respiration rate returned to normal indicating that the above changes are reversible In a longitudinal study, the effects of cholecalciferol therapy on skeletal mitochondrial oxidative function in vitamin D deficient subjects using 31Phosphorus magnetic resonance spectroscopy were examined.The phosphocreatine recovery half-time (t1/2PCr) was significantly reduced after cholecalciferol therapy in the subjects indicating an improvement in maximal oxidative phosphorylation (34.44 ±8.18 sec to 27.84 ±9.54 sec, P <.001).

Thus, vitamin D may improve the statin-mediated changes in cardiorespiratory fitness and mitochondrial function by improving the enzymatic machinery involved in oxidative phosphorylation which is blocked by statin. Another proposed mechanism of interaction between statin and vitamin D is inhibition of CYP3A4 by statins, which displays 25-hydroxylase activity in vitro. Vitamin D deficiency leads to 'preferential shunting' of CYP3A4 for hydroxylation of vitamin D, thus decreasing the availability of CYP3A4 for statin metabolism leading to statin-induced toxicity.

This study describes the effect of vitamin D supplementation on simvastatin-mediated change in exercise-mediated cardiorespiratory fitness and skeletal muscle mitochondrial content in adults with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes Mellitus
* No significant microvascular complication
* Age between 25 and 50 yrs
* HbA1c<7.5%
* LDL-C between 100 to 130mg/dl
* Overweight or obese (BMI 25 -39 kg/m2)
* Low physical activity(WHO-GPAQ)
* Euthyroid , Eugonadal
* Vitamin D deficient (<20 ng/ml)
* Normal ECG

Exclusion Criteria:

* Use of statins in past 3 months
* Use of Thiazolidinediones, Glucagon like peptide -1agonists, Dipeptidyl Peptidase -IV inhibitors, steroids, orlistat or other medicines affecting lipid profile or body weight
* Smoking
* On Vitamin D supplementation
* Uncontrolled DM with HbA1c>7.5
* Uncontrolled hypertension
* Significant microvascular complication of DM
* Macrovascular disease
* Musculoskeletal problems resulting in inability to exercise
* Pregnancy

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil Bhansali, DM, Principal Investigator — PGIMER, Chandigarh
Locations (1):
- PGIMER, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Simvastatin and Placebo: Eleven participants will be vitamin D deficient with LDL-C between 100 to 130mg/dl This arm will receive simvastatin 40 mg once daily and placebo once weekly , and will exercise for twelve weeks
- Simvastatin and Vitamin D: Eleven participants will be vitamin D deficient with LDL-C between 100 to 130mg/dl This arm will receive Simvastatin 40 mg once daily and vitamin D 60000 units once weekly, and will exercise for twelve weeks
- Vitamin D and Placebo: Eleven participants will be vitamin D deficient with LDL-C between 100 to 130mg/dl This arm will receive vitamin D 60,000 units once weekly and placebo once daily, and will exercise for twelve weeks
Period: Overall Study
Arm/Group | Simvastatin and Placebo | Simvastatin and Vitamin D | Vitamin D and Placebo
Started | 11 | 11 | 11
Completed | 9 | 9 | 10
Not Completed | 2 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Simvastatin and Placebo: Participants took simvastatin 40 mg once daily and performed exercise for 12 weeks
- Simvastatin and Vitamin D: Participants took simvastatin 40 mg once daily and vitamin D 60,000 units once weekly, and performed exercise for 12 weeks
- Vitamin D and Placebo: Participants took vitamin D 60000 units once weekly and performed exercise for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Simvastatin and Placebo | Simvastatin and Vitamin D | Vitamin D and Placebo | Total
Number analyzed (Participants) | 9 | 9 | 10 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 10 | 28
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 5
  Male | 8 | 6 | 9 | 23
Race/Ethnicity, Customized [Number; unit: participants]
  Asian Indian | 9 | 9 | 10 | 28
Region of Enrollment [Number; unit: participants]
  India | 9 | 9 | 10 | 28
Body mass index(BMI) [Mean (Standard Deviation); unit: kg/m2] | 27.9 (2.4) | 28.1 (2.5) | 27.4 (2.2) | 27.8 (2.4)
HbA1c [Mean (Standard Deviation); unit: %] | 6.9 (0.4) | 6.9 (0.5) | 6.9 (0.5) | 6.9 (0.5)
Fasting plasma Insulin [Mean (Standard Deviation); unit: microIU/ml] | 13.6 (6.3) | 12.1 (5) | 13.2 (4.5) | 13.1 (5.2)
Low density Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mg/dl] | 117.4 (9.4) | 116.4 (11.4) | 112 (6.8) | 115.2 (9.3)
Peak oxygen consumption(VO2peak) [Mean (Standard Deviation); unit: L/min] — Peak oxygen consumption (VO2peak) is defined as highest rate at which oxygen can be taken up and utilized by body during severe exercise during bicycle ergometry The participants were encouraged to exercise to exhaustion with progressive 2-minutes increments in the power output during the test. VO2peak was obtained when participants reached volitional exhaustion and met one of the following criteria: plateau in oxygen consumption despite increase in workload, rating of perceived exertion >18, Respiratory exchange ratio > 1.10 and peak heart rate within 10 beats of age predicted maximum.
  L/min | 1.33 (0.5) | 1.13 (0.4) | 1.1 (0.2) | 1.2 (0.4)
Peak oxygen consumption percentage of predicted value (VO2peak%) [Mean (Standard Deviation); unit: %] — As VO2peak (expressed as liters of oxygen consumed per minute) is also dependent on age, sex, and body size, it was also expressed as percentage of the predicted value(VO2peak%).
  % | 52.2 (9.8) | 52.2 (8.9) | 46.4 (8.6) | 50.1 (9.2)
Skeletal muscle citrate synthase activity [Mean (Standard Deviation); unit: change in mOD/min at 412nm] — Skeletal muscle citrate synthase activity is a validated marker of mitochondrial content.Skeletal muscle biopsy is obtained from vastus lateralis muscle of five patients in either groups before and after the intervention. Under aseptic conditions, samples were taken in protease inhibitor cocktail and stored at -80ºcelsius. Mitochondrial citrate synthase activity (the working range of the kit was 1.56-100 µg/mL, with intra and inter assay coefficient of variation (CV) of 4.35-6.55 % and 8.3 % respectively) is measured using ELISA Kit (Abcam, Cambridge, UK) as per manufacturer's instructions.
  change in mOD/min at 412nm | 0.0051 (0.0001) | 0.0042 (0.0019) | 0.0043 (0.0017) | 0.0046 (0.0013)

OUTCOME MEASURES:

1. Primary Outcome: Peak Oxygen Consumption
Description: Peak oxygen consumption( VO2peak) is defined as the highest rate at which oxygen can be taken up and utilized by the body during severe exercise. The participants were encouraged to exercise to exhaustion with progressive 2-minutes increments in the power output during the test. VO2peak was obtained when participants reached volitional exhaustion and met at least one of the following criteria: plateau in oxygen consumption despite increase in workload, rating of perceived exertion >18, Respiratory exchange ratio > 1.10 and peak heart rate within 10 beats of age predicted maximum. . As VO2peak (expressed as liters of oxygen consumed per minute) is also dependent on age, sex, and body size, it was expressed as percentage of the predicted value(VO2peak%).
Time Frame: Twelve weeks
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Groups:
- Simvastatin and Placebo: Participants received simvastatin 40 mg once daily and performed exercise for 12 weeks
- Simvastatin and Vitamin D: Participants received simvastatin 40 mg once daily and vitamin D 60,000 units once weekly, and performed exercise for 12 weeks
- Vitamin D and Placebo: Participants received vitamin D 60,000 units once weekly and performed exercise for 12 weeks
Arm/Group | Simvastatin and Placebo | Simvastatin and Vitamin D | Vitamin D and Placebo
Number analyzed (Participants) | 9 | 9 | 10
percentage of predicted value | 43.8 (7.3) | 51.6 (10.5) | 53.5 (10.4)

2. Primary Outcome: Skeletal Muscle Mitochondrial Content
Description: Skeletal muscle citrate synthase activity is a validated marker of mitochondrial content. Skeletal muscle biopsy was obtained from vastus lateralis muscle of five patients in either groups before and after the intervention. Under aseptic conditions, samples were taken in protease inhibitor cocktail and stored at -80ºC. Mitochondrial citrate synthase activity (the working range of the kit was 1.56-100 µg/mL, with intra and inter assay CV of 4.35-6.55 % and 8.3 % respectively) was measured using ELISA Kit (Abcam, Cambridge, UK) as per manufacturer's instructions.Skeletal muscle citrate synthase activity is a validated marker of mitochondrial content.
Time Frame: Twelve weeks
Measure: Mean (Standard Deviation); unit: change in mOD/min at 412nm
Arm/Group | Simvastatin and Placebo | Simvastatin and Vitamin D | Vitamin D and Placebo
Number analyzed (Participants) | 9 | 9 | 10
change in mOD/min at 412nm | 0.005 (0.0007) | 0.005 (0.0001) | 0.0052 (0.0001)

ADVERSE EVENTS:
Groups:
- Simvastatin and Placebo: Eleven participants will be vitaminD deficient with LDL-C between 100 to 130mg/dl This arm will receive Simvastatin 40 mg once daily and placebo once weekly, and will exercise for twelve weeks
  Simvastatin: Simvastatin in a dose of 40 mg will be provided to the study participants
  Placebo: Placebo will be provided to the study participants
- Simvastatin and Vitamin D: Eleven participants will be vitamin D deficient with LDL-C between 100 to 130mg/dl This arm will receive simvastatin 40 mg once daily and vitamin D 60,000 units once weekly , and will exercise for twelve weeks
  Vitamin D: Vitamin D will be given to achieve normal serum levels
  Simvastatin: Simvastatin in a dose of 40 mg will be provided to the study participants
Arm/Group | Simvastatin and Placebo | Simvastatin and Vitamin D | Vitamin D and Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 2/9 | 1/9 | 0/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simvastatin and Placebo (N=9) | Simvastatin and Vitamin D (N=9) | Vitamin D and Placebo (N=10)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0

LIMITATIONS AND CAVEATS:
The limitations include short duration of follow up and lack of direct supervision of exercise program. Although participants didn't perform exercise under direct supervision, adherence to exercise program was monitored by pedometer readings weekly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes